CLINICAL TRIAL: NCT01944800
Title: Prospective, Randomized Trial of Ticagrelor Versus Prasugrel in Patients With Acute Coronary Syndrome - Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 5
Brief Title: Prospective, Randomized Trial of Ticagrelor Versus Prasugrel in Patients With Acute Coronary Syndrome
Acronym: ISAR-REACT 5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE 00113; 2013-002272-40 (EudraCT Number)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Ticagrelor; Prasugrel; Acute coronary syndrome; Percutaneous coronary intervention
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- Prasugrel (Active Comparator)
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Ticagrelor — Loading dose of 180 mg, followed by maintenance dose of 180 mg per day
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Prasugrel — Loading dose of 60 mg, followed by maintenance dose of 10 mg/day or 5 mg/day in patients =/> 75 years or < 60 kg
  Other Names: Efient
  Arms: Prasugrel

SUMMARY:
Aim of the randomized, open-label, multicenter ISAR-REACT 5 trial is to assess whether ticagrelor is superior to prasugrel in patients with acute coronary syndrome and planned invasive strategy in terms of clinical outcomes.

ELIGIBILITY:
Major Inclusion Criteria:

Hospitalization for an acute coronary syndrome (ST-segment elevation myocardial infarction, non-ST-segment elevation myocardial infarction or unstable angina pectoris) with planned invasive strategy

Major Exclusion Criteria:

1. intolerance of or allergy to ticagrelor or prasugrel
2. history of any stroke, transient ischemic attack or intracranial bleeding
3. known intracranial neoplasm, intracranial arteriovenous malformation or intracranial aneurysm
4. active bleeding, clinical findings, that in the judgement of the investigator are associated with an increased risk of bleeding
5. fibrin-specific fibrinolytic therapy less than 24 h before randomization, non-fibrin-specific fibrinolytic therapy less than 48 h before randomization
6. known platelet count < 100.000/μL at the time of screening
7. known anemia (hemoglobin <10 g/dL) at the time of screening
8. oral anticoagulation that cannot be safely discontinued for the duration of the study
9. INR known to be greater than 1.5 at the time of screening
10. chronic renal insufficiency requiring dialysis
11. moderate or severe hepatic dysfunction (Child Pugh B or C)
12. increased risk of bradycardia events (Sick Sinus, AV block grade II or III, bradycardia-induced syncope)
13. index event is an acute complication (< 30 days) of PCI
14. concomitant medical illness that in the opinion of the investigator is associated with a life expectancy < 1 year
15. concomitant oral or i.v. therapy with strong CYP3A Inhibitors (e.g. ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice > 1 L/d), CYP3A substrates with narrow therapeutic indices (e.g. cyclosporine, quinidine), or strong CYP3A inducers (e.g. rifampin/rifampicin, phenytoin, carbamazepine, dexamethason, phenobarbital ) that cannot be safely discontinued
16. ≥1 doses of ticagrelor or prasugrel within 5 days before randomisation
17. no written informed consent
18. participation in another investigational drug study
19. previous enrolment in this study
20. for women of childbearing potential no negative pregnancy test and no agree to use reliable method of birth control during the study
21. Pregnancy, giving birth within the last 90 days, or lactation
22. inability to cooperate with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4018 (Actual)
Dates: Start 2013-09-15 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Composite of death, myocardial infarction or stroke | 12 months

SECONDARY OUTCOMES:
Bleeding | 12 months
  Bleeding according to BARC
Mortality | 12 months
  Death for any cause
Stroke | 12 months
  Stroke
Myocardial Infarction | 12 months
Stent Thrombosis | 12 months
  Stent thrombosis according to ARC

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum München; Stefanie Schuepke, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (19):
- Germany (17):
  - Universitäts-Herzzentrum Freiburg/ Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Universitäts-Klinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Landkreis Erding, Erding, Bavaria
  - Deutsches Herzzentrum Munich, München, Bavaria
  - Klinikum rechts der Isar, 1. Medizinische Klinik und Poliklinik, München, Bavaria
  - Klinikum Neuperlach, München, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Klinikum Traunstein, Traunstein, Bavaria
  - Kerckhoff-Klinik GmbH, Abteilung für Kardiologie, Bad Nauheim, Hesse
  - Universitätsmedizin Göttingen, Herzzentrum, Göttingen, Lower Saxony
  - Herzzentrum Wuppertal, Wuppertal, North Rhine-Westphalia
  - Segeberger Kliniken GmbH, Bad Segeberg, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Klinik für Innere Medizin III, Campus Kiel, Kiel, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Charité Universitätsmedizin Berlin, Campus Virchow-Klinik, Berlin
- Italy (2):
  - Careggi University Hospital, Invasive Cardiology Division, Florence
  - Spaziani Hospital Frosinone, Frosinone

REFERENCES:
- [Derived] Bongiovanni D, Schreiner N, Gosetti R, Mayer K, Angiolillo DJ, Sibbing D, Holdenrieder S, Anetsberger A, von Scheidt M, Schunkert H, Laugwitz KL, Schupke S, Kastrati A, Fegers-Wustrow I, Bernlochner I. Immature Platelet Fraction Predicts Adverse Events in Patients With Acute Coronary Syndrome: the ISAR-REACT 5 Reticulated Platelet Substudy. Arterioscler Thromb Vasc Biol. 2023 Feb;43(2):e83-e93. doi: 10.1161/ATVBAHA.122.318614. Epub 2022 Dec 22. PMID 36546322
- [Derived] Lahu S, Scalamogna M, Ndrepepa G, Menichelli M, Valina C, Hemetsberger R, Witzenbichler B, Bernlochner I, Joner M, Xhepa E, Hapfelmeier A, Kufner S, Sager HB, Mayer K, Kessler T, Laugwitz KL, Richardt G, Schunkert H, Neumann FJ, Kastrati A, Cassese S. Prior Myocardial Infarction and Treatment Effect of Ticagrelor Versus Prasugrel in Patients With Acute Coronary Syndromes - A Post-hoc Analysis of the ISAR-REACT 5 Trial. J Am Heart Assoc. 2022 Dec 20;11(24):e027257. doi: 10.1161/JAHA.122.027257. Epub 2022 Dec 14. PMID 36515247
- [Derived] Aytekin A, Coughlan JJ, Ndrepepa G, Cassese S, Lahu S, Kufner S, Mayer K, Xhepa E, Gewalt S, Joner M, Hapfelmeier A, Angiolillo DJ, Menichelli M, Richardt G, Neumann FJ, Schunkert H, Kastrati A. The effect of a Prasugrel- vs. a Ticagrelor-based strategy on total ischaemic and bleeding events in patients with acute coronary syndromes. Eur Heart J Cardiovasc Pharmacother. 2023 Apr 10;9(3):231-239. doi: 10.1093/ehjcvp/pvac067. PMID 36434779
- [Derived] Lahu S, Presch A, Ndrepepa G, Menichelli M, Valina C, Hemetsberger R, Witzenbichler B, Bernlochner I, Joner M, Xhepa E, Hapfelmeier A, Kufner S, Rifatov N, Sager HB, Mayer K, Kessler T, Laugwitz KL, Richardt G, Schunkert H, Neumann FJ, Sibbing D, Angiolillo DJ, Kastrati A, Cassese S. Ticagrelor or Prasugrel in Patients With Acute Coronary Syndrome and High Bleeding Risk. Circ Cardiovasc Interv. 2022 Oct;15(10):e012204. doi: 10.1161/CIRCINTERVENTIONS.122.012204. Epub 2022 Oct 18. PMID 36256695
- [Derived] Behnes M, Lahu S, Ndrepepa G, Menichelli M, Mayer K, Wohrle J, Bernlochner I, Gewalt S, Witzenbichler B, Hochholzer W, Sibbing D, Cassese S, Angiolillo DJ, Hemetsberger R, Valina C, Muller A, Kufner S, Hamm CW, Xhepa E, Hapfelmeier A, Sager HB, Joner M, Fusaro M, Richardt G, Laugwitz KL, Neumann FJ, Schunkert H, Schupke S, Kastrati A, Akin I. Ticagrelor or prasugrel in patients with acute coronary syndrome with off-hour versus on-hour presentation: a subgroup analysis of the ISAR-REACT 5 trial. Clin Res Cardiol. 2023 Apr;112(4):518-528. doi: 10.1007/s00392-022-02040-z. Epub 2022 Jul 5. PMID 35789430
- [Derived] Hemetsberger R, Richardt G, Lahu S, Valina C, Menichelli M, Abdelghani M, Wohrle J, Toelg R, Witzenbichler B, Mankerious N, Liebetrau C, Bernlochner I, Hamm CW, Allali A, Joner M, Fusaro M, Xhepa E, Hapfelmeier A, Kufner S, Sager HB, Schupke S, Laugwitz KL, Schunkert H, Neumann FJ, Kastrati A, Cassese S. Access Route and Clinical Outcomes After Ticagrelor Versus Prasugrel in Patients With Acute Coronary Syndrome Undergoing Invasive Treatment Strategy. Cardiovasc Revasc Med. 2022 Aug;41:122-128. doi: 10.1016/j.carrev.2021.12.029. Epub 2022 Jan 3. PMID 35045943
- [Derived] Lahu S, Behnes M, Ndrepepa G, Neumann FJ, Sibbing D, Bernlochner I, Menichelli M, Mayer K, Richardt G, Gewalt S, Angiolillo DJ, Coughlan JJ, Aytekin A, Witzenbichler B, Hochholzer W, Cassese S, Kufner S, Xhepa E, Sager HB, Joner M, Fusaro M, Laugwitz KL, Schunkert H, Schupke S, Kastrati A, Akin I. Body mass index and efficacy and safety of ticagrelor versus prasugrel in patients with acute coronary syndromes. Rev Esp Cardiol (Engl Ed). 2022 Sep;75(9):747-755. doi: 10.1016/j.rec.2021.11.007. Epub 2021 Dec 24. English, Spanish. PMID 34961732
- [Derived] Ndrepepa G, Neumann FJ, Menichelli M, Bernlochner I, Richardt G, Wohrle J, Witzenbichler B, Mayer K, Cassese S, Gewalt S, Xhepa E, Kufner S, Sager HB, Joner M, Ibrahim T, Laugwitz KL, Schunkert H, Schupke S, Kastrati A. Assessment of Impact of Patient Recruitment Volume on Risk Profile, Outcomes, and Treatment Effect in a Randomized Trial of Ticagrelor Versus Prasugrel in Acute Coronary Syndromes. J Am Heart Assoc. 2021 Nov 16;10(22):e021418. doi: 10.1161/JAHA.121.021418. Epub 2021 Nov 15. PMID 34779234
- [Derived] Ndrepepa G, Holdenrieder S, Neumann FJ, Lahu S, Cassese S, Joner M, Xhepa E, Kufner S, Wiebe J, Laugwitz KL, Gewalt S, Schunkert H, Kastrati A. Prognostic value of glomerular function estimated by Cockcroft-Gault creatinine clearance, MDRD-4, CKD-EPI and European Kidney Function Consortium equations in patients with acute coronary syndromes. Clin Chim Acta. 2021 Dec;523:106-113. doi: 10.1016/j.cca.2021.09.007. Epub 2021 Sep 13. PMID 34529983
- [Derived] Coughlan JJ, Aytekin A, Ndrepepa G, Schupke S, Bernlochner I, Mayer K, Neumann FJ, Menichelli M, Richardt G, Wohrle J, Xhepa E, Kufner S, Sager HB, Joner M, Ibrahim T, Fusaro M, Laugwitz KL, Schunkert H, Kastrati A, Cassese S. Twelve-month clinical outcomes in patients with acute coronary syndrome undergoing complex percutaneous coronary intervention: insights from the ISAR-REACT 5 trial. Eur Heart J Acute Cardiovasc Care. 2021 Dec 18;10(10):1117-1124. doi: 10.1093/ehjacc/zuab077. PMID 34468709
- [Derived] Wohrle J, Seeger J, Lahu S, Mayer K, Bernlochner I, Gewalt S, Menichelli M, Witzenbichler B, Hochholzer W, Sibbing D, Cassese S, Angiolillo DJ, Hemetsberger R, Valina C, Kufner S, Xhepa E, Hapfelmeier A, Sager HB, Joner M, Richardt G, Laugwitz KL, Neumann FJ, Schunkert H, Schupke S, Kastrati A, Ndrepepa G. Ticagrelor or Prasugrel in Patients With Acute Coronary Syndrome in Relation to Estimated Glomerular Filtration Rate. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1857-1866. doi: 10.1016/j.jcin.2021.06.028. Epub 2021 Aug 23. PMID 34446390
- [Derived] Coughlan JJ, Aytekin A, Lahu S, Ndrepepa G, Menichelli M, Mayer K, Wohrle J, Bernlochner I, Gewalt S, Witzenbichler B, Hochholzer W, Sibbing D, Cassese S, Angiolillo DJ, Hemetsberger R, Valina C, Muller A, Kufner S, Liebetrau C, Xhepa E, Hapfelmeier A, Sager HB, Joner M, Fusaro M, Richardt G, Laugwitz KL, Neumann FJ, Schunkert H, Schupke S, Kastrati A. Ticagrelor or Prasugrel for Patients With Acute Coronary Syndrome Treated With Percutaneous Coronary Intervention: A Prespecified Subgroup Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2021 Oct 1;6(10):1121-1129. doi: 10.1001/jamacardio.2021.2228. PMID 34190967
- [Derived] Coughlan JJ, Aytekin A, Ndrepepa G, Schupke S, Bernlochner I, Mayer K, Neumann FJ, Menichelli M, Richardt G, Wohrle J, Witzenbichler B, Gewalt S, Xhepa E, Kufner S, Sager HB, Joner M, Ibrahim T, Fusaro M, Laugwitz KL, Schunkert H, Kastrati A, Cassese S. Ticagrelor or Prasugrel in Patients With Acute Coronary Syndrome Undergoing Complex Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2021 Jul;14(7):e010565. doi: 10.1161/CIRCINTERVENTIONS.121.010565. Epub 2021 Jun 16. PMID 34130477
- [Derived] Lahu S, Ndrepepa G, Gewalt S, Schupke S, Pellegrini C, Bernlochner I, Aytekin A, Neumann FJ, Menichelli M, Richardt G, Cassese S, Xhepa E, Kufner S, Sager HB, Joner M, Ibrahim T, Fusaro M, Laugwitz KL, Schunkert H, Kastrati A, Mayer K. Efficacy and safety of ticagrelor versus prasugrel in smokers and nonsmokers with acute coronary syndromes. Int J Cardiol. 2021 Sep 1;338:8-13. doi: 10.1016/j.ijcard.2021.06.011. Epub 2021 Jun 11. PMID 34126130
- [Derived] Mayer K, Bongiovanni D, Karschin V, Sibbing D, Angiolillo DJ, Schunkert H, Laugwitz KL, Schupke S, Kastrati A, Bernlochner I. Ticagrelor or Prasugrel for Platelet Inhibition in Acute Coronary Syndrome Patients: The ISAR-REACT 5 Trial. J Am Coll Cardiol. 2020 Nov 24;76(21):2569-2571. doi: 10.1016/j.jacc.2020.09.586. No abstract available. PMID 33213734
- [Derived] Valina C, Neumann FJ, Menichelli M, Mayer K, Wohrle J, Bernlochner I, Aytekin A, Richardt G, Witzenbichler B, Sibbing D, Cassese S, Angiolillo DJ, Kufner S, Liebetrau C, Hamm CW, Xhepa E, Hapfelmeier A, Sager HB, Wustrow I, Joner M, Trenk D, Laugwitz KL, Schunkert H, Schupke S, Kastrati A. Ticagrelor or Prasugrel in Patients With Non-ST-Segment Elevation Acute Coronary Syndromes. J Am Coll Cardiol. 2020 Nov 24;76(21):2436-2446. doi: 10.1016/j.jacc.2020.09.584. PMID 33213722
- [Derived] Aytekin A, Ndrepepa G, Neumann FJ, Menichelli M, Mayer K, Wohrle J, Bernlochner I, Lahu S, Richardt G, Witzenbichler B, Sibbing D, Cassese S, Angiolillo DJ, Valina C, Kufner S, Liebetrau C, Hamm CW, Xhepa E, Hapfelmeier A, Sager HB, Wustrow I, Joner M, Trenk D, Fusaro M, Laugwitz KL, Schunkert H, Schupke S, Kastrati A. Ticagrelor or Prasugrel in Patients With ST-Segment-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention. Circulation. 2020 Dec 15;142(24):2329-2337. doi: 10.1161/CIRCULATIONAHA.120.050244. Epub 2020 Oct 29. PMID 33115278
- [Derived] Ndrepepa G, Kastrati A, Menichelli M, Neumann FJ, Wohrle J, Bernlochner I, Richardt G, Witzenbichler B, Sibbing D, Gewalt S, Angiolillo DJ, Hamm CW, Hapfelmeier A, Trenk D, Laugwitz KL, Schunkert H, Schupke S, Mayer K. Ticagrelor or Prasugrel in Patients With Acute Coronary Syndromes and Diabetes Mellitus. JACC Cardiovasc Interv. 2020 Oct 12;13(19):2238-2247. doi: 10.1016/j.jcin.2020.07.032. PMID 33032712
- [Derived] Menichelli M, Neumann FJ, Ndrepepa G, Mayer K, Wohrle J, Bernlochner I, Richardt G, Witzenbichler B, Sibbing D, Gewalt S, Angiolillo DJ, Lahu S, Hamm CW, Hapfelmeier A, Trenk D, Laugwitz KL, Schunkert H, Schupke S, Kastrati A. Age- and Weight-Adapted Dose of Prasugrel Versus Standard Dose of Ticagrelor in Patients With Acute Coronary Syndromes : Results From a Randomized Trial. Ann Intern Med. 2020 Sep 15;173(6):436-444. doi: 10.7326/M20-1806. Epub 2020 Jul 21. PMID 32687741
- [Derived] Schupke S, Neumann FJ, Menichelli M, Mayer K, Bernlochner I, Wohrle J, Richardt G, Liebetrau C, Witzenbichler B, Antoniucci D, Akin I, Bott-Flugel L, Fischer M, Landmesser U, Katus HA, Sibbing D, Seyfarth M, Janisch M, Boncompagni D, Hilz R, Rottbauer W, Okrojek R, Mollmann H, Hochholzer W, Migliorini A, Cassese S, Mollo P, Xhepa E, Kufner S, Strehle A, Leggewie S, Allali A, Ndrepepa G, Schuhlen H, Angiolillo DJ, Hamm CW, Hapfelmeier A, Tolg R, Trenk D, Schunkert H, Laugwitz KL, Kastrati A; ISAR-REACT 5 Trial Investigators. Ticagrelor or Prasugrel in Patients with Acute Coronary Syndromes. N Engl J Med. 2019 Oct 17;381(16):1524-1534. doi: 10.1056/NEJMoa1908973. Epub 2019 Sep 1. PMID 31475799
- [Derived] Schulz S, Angiolillo DJ, Antoniucci D, Bernlochner I, Hamm C, Jaitner J, Laugwitz KL, Mayer K, von Merzljak B, Morath T, Neumann FJ, Richardt G, Ruf J, Schomig G, Schuhlen H, Schunkert H, Kastrati A; Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 5 Trial Investigators. Randomized comparison of ticagrelor versus prasugrel in patients with acute coronary syndrome and planned invasive strategy--design and rationale of the iNtracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 5 trial. J Cardiovasc Transl Res. 2014 Feb;7(1):91-100. doi: 10.1007/s12265-013-9527-3. Epub 2013 Dec 27. PMID 24371012